CLINICAL TRIAL: NCT05254366
Title: A Domestic, Prospective, Non-interventional Study of Remazolam Methyl Benzene Sulfonic Acid for Injection in Real-world Clinical Practice
Brief Title: A Non-interventional Study of Remazolam Methyl Benzene Sulfonic Acid for Injection in Real-world Clinical Practice
Status: Completed | Type: Observational
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: ARMS
Record Dates: First submitted 2022-01-28; First posted 2022-02-24 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Gastroscopic and Colonoscopic Sedation
MeSH Terms: interventions — Injections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Painless gastroscopic sedation cohort
  Interventions: Drug: Remimazolam Tosilate for Injection
- Cohort 2: Painless colonoscopy sedation cohort
  Interventions: Drug: Remimazolam Tosilate for Injection

INTERVENTIONS:
Drug: Remimazolam Tosilate for Injection — Remimazolam Tosilate for Injection

SUMMARY:
This is a non-interventional study of remazolam toluenesulfonate (rebenin ®) for injection in Chinese patients. A total of 2000 patients were enrolled in this study based on the preliminary safety assessment of rebenin ®, and all safety information was obtained

ELIGIBILITY:
Inclusion Criteria:

1. Use rebenin ® for painless gastroscopic sedation and painless colonoscopic sedation
2. Patients need to sign informed consent

Exclusion Criteria:

1. Patients who are participating in or planning to participate in any interventional clinical trial
2. The investigator considers that there are any other reasons for the patient's ineligibility for the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients receiving remazolam toluenesulfonate for painless gastroscopy and colonoscopy
Sampling Method: Non-Probability Sample
Enrollment: 2022 (Actual)
Dates: Start 2022-01-30 (Actual); Primary Completion 2023-02-08 (Actual); Study Completion 2023-02-08 (Actual)

PRIMARY OUTCOMES:
Adverse events | Within 3 days of receiving gastroscopy and colonoscopy
  Use adverse event record form,Refer to version 5.0 of the NCI-CTCAE

SECONDARY OUTCOMES:
Serious adverse events | Within 3 days of receiving gastroscopy and colonoscopy
  Refer to SAE definition standards
Adverse drug reactions | Within 3 days of receiving gastroscopy and colonoscopy
  By evaluating the association of adverse events with drugs
Injection pain questionnaire | Within 3 days of receiving gastroscopy and colonoscopy
  By observing and asking

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided